CLINICAL TRIAL: NCT06673264
Title: FINESSE: First-In-Human Trial Using a NovEl Soft Neural Probe: an IDEAL StagE 1 Study
Brief Title: First-In-human Trial of a NovEl Soft and Stretchable Neural probE
Acronym: FINESSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axoft, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PLAN-000045
Record Dates: First submitted 2024-10-25; First posted 2024-11-04 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Feasibility of Safe Insertion and Neural Recording With a Soft Neural Probe; Brain Surgery
Keywords: First-in-human; Brain-Computer Interface

STUDY DESIGN:
Intervention Model Description: Participants undergoing brain resection due to tumor or epilepsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Receives soft neural probe device insertion (Experimental)
  Interventions: Device: Soft Neural Probe

INTERVENTIONS:
Device: Soft Neural Probe — sub-acute insertion of the soft neural probe with neural signal recording

SUMMARY:
The goal of this interventional study is to find out the feasibility of whether the soft neural probe can be used in human brain tissue. The main questions it aims to answer are:

* Are there any problems when inserting the soft neural probe into brain tissue?
* Can the soft neural probe record electrical signals from the brain tissue?

Participants will:

* During their already scheduled brain tumor or epileptic tissue removal, have the soft neural probe inserted into the section of brain tissue that is due to be removed
* Visit the clinic for follow up after 30 days for checkups

ELIGIBILITY:
Inclusion Criteria

* Adults 18-80 years of age at the time of providing informed consent
* Capable of providing written informed consent to participate
* Willing to commit to the study evaluations and visit schedule
* Undergoing a planned surgery for brain tissue resection of either a tumor or of a epileptogenic lesion
* Adequate hepatic, renal, cardiac, and hematologic function according to the following laboratory test criteria:

  * Absolute neutrophil count ≥ 1,500/mm3
  * Platelet count ≥ 100,000/mm3
  * Bilirubin ≤ 1.5 mg/dL
  * AST and ALT ≤ 2.5 times upper limit of normal
  * Creatinine ≤ 1.5 mg/dL
  * Signs of previous or current ischemic cardiac disease or arrhythmia per electrocardiogram assessment
* Females of childbearing potential must have a negative serum pregnancy test and agree to use birth control measures during study treatment and for 3 months after its completion
* Must not be pregnant or nursing at study entry
* Women/men of reproductive potential must have agreed to use an effective contraceptive method

Exclusion Criteria

* Substance abuse, according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5)
* Allergy to any study materials
* Presence of any powered implantable medical device or any medical device implanted in the brain
* Weakened immune system due to presence of poorly controlled chronic diseases such as human immunodeficiency virus (seropositive for HIV 1 or 2), decompensated diabetes, decompensated chronic kidney disease, decompensated liver disease, intake of immunosuppressive medications such as high-dose corticosteroids, or a previous diagnosis of congenital or acquired immunodeficiency
* Exposure to any type of chemotherapy in the past 3 months
* Radiation therapy in the surgical area within the last year
* Delay to the base operation creates additional risk for the patient due to uncontrolled elevated ICP or emergency surgery
* Active infection, bleeding, or hematoma
* Patients with previous resection surgery in the planned surgical area
* Previous stroke in the affected tissue
* Currently high levels of inflammation as indicated by ESR, CRP, or PCT blood test
* Any concurrent medical condition or disease (e.g. uncontrolled active hypertension, uncontrolled active diabetes, or active systemic infection) that is likely to interfere with study procedures.
* Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 1 week prior to the planned neurosurgical intervention. Patients on prophylactic antibiotics or with a controlled infection within 1 week prior to the planned neurosurgical intervention are acceptable.
* Any active, serious psychiatric, medical, or other conditions/situations that, in the opinion of the Investigator, could interfere with treatment, compliance, or the ability to give informed consent.
* Any other psychological, family or geographic problem that may make compliance with the study protocol difficult.
* Life expectancy of less than 3 months.
* Major surgery within 4 weeks prior to planned neurosurgical intervention

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed by adverse events | From surgery to 30-day follow up
  Assessed by enumerating reported adverse events occurring from use of the study device during the study period.

SECONDARY OUTCOMES:
Feasibility assessed by use | From the introduction of the soft neural probe into the surgery field until 20 minutes later
  Assessed by average of Net Promoter Score
Local tissue effect biocompatibility via measurement of area of affected tissue | Histopathology conducted within 3 months following tissue resection
  Histopathological evaluation of the resected tissue including the insertion track of the soft neural probe. Area of tissue damaged as defined by H&E staining
Number of Participants where Neural Signals are Recorded from the Soft Neural Probe | From the introduction of the soft neural probe into the surgery field until 20 minutes later

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Vacunación e Investigación SA (CEVAXIN) - The Panama Clinic, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No